CLINICAL TRIAL: NCT00606840
Title: Study to Prevent Weight Gain
Brief Title: Weight Gain Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Jessica LaRose, Assistant Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #2018-07
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Weight Gain
Keywords: overweight; prevention of weight gain; young adults; self-regulation; daily weighing; weight gain prevention
MeSH Terms: conditions — Weight Gain; Overweight; Self-Control | interventions — Eating; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): One arm is a large changes group in which participants will be asked to make periodic large changes in their eating and activity, aimed at producing initial weight loss, in order to prevent weight gain over time.
  Interventions: Behavioral: large changes in eating and activity
- 2 (Experimental): The second arm is a small changes group in which participants will be asked to make small changes to their eating and activity and maintain these changes forever in order to prevent weight gain.
  Interventions: Behavioral: small changes in eating and activity

INTERVENTIONS:
Behavioral: large changes in eating and activity — Behavioral self-regulation interventions to prevent weight gain in young adults.
  Arms: 1
Behavioral: small changes in eating and activity — Behavioral self-regulation interventions to prevent weight gain in young adults.
  Arms: 2

SUMMARY:
The specific aim of the proposed project is to test two separate self-regulation interventions to prevent weight gain in young adults, one based on making sustained small changes in behavior to prevent weight gain and the other on making periodic larger behavior changes resulting in weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Body mass index between 23 and 30
* Interested in preventing weight gain

Exclusion Criteria:

* BMI outside of range specified
* Age outside of range specified
* History of or current eating disorder or substance abuse
* Recent weight loss greater than 5% of weight
* Currently in another research study that would interfere

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
weight change | 8 weeks and 16 weeks

SECONDARY OUTCOMES:
frequency of weighing, adherence to intervention, diet, activity | 8 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States